CLINICAL TRIAL: NCT05386290
Title: A Multicentered Prospective Cohort Study of Chinese IBD Patients Concerning Cost-effectiveness Analysis, Therapeutic Effect Predictor Exploration and Gut Microbiota Analysis
Brief Title: A Multicentered Prospective Cohort Study of Chinese IBD Patients
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Hong Yang, Professor, Peking Union Medical College Hospital
Other Study IDs: JS-3086
Record Dates: First submitted 2022-05-17; First posted 2022-05-23 (Actual); Last update posted 2022-05-23 (Actual); Status verified 2022-05

CONDITIONS: Ulcerative Colitis; Crohn Disease
MeSH Terms: conditions — Colitis, Ulcerative; Crohn Disease | interventions — Infliximab; vedolizumab; Ustekinumab; Mesalamine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Patients' residual blood sample after test and stool specimen are collected.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- UC patients: Patients who were diagnosed moderate-to-severe ulcerative colitis (UC) and intend to be treated by biological agents (infliximab or vedolizumab) or traditional drugs (glucocoticoid, immunosupressive drugs and/or mesalazine) will be enrolled.
  Interventions: Drug: Infliximab; Drug: Vedolizumab; Drug: conventional treatment (glucocoticoid, immunosupressive drugs and/or mesalazine)
- CD patients: Patients who were diagnosed moderate-to-severe Crohn's Disease (CD) and intend to be treated by biological agents (infliximab or ustekinumab) or traditional drugs (glucocoticoid, immunosupressive drugs and/or mesalazine) will be enrolled.
  Interventions: Drug: Infliximab; Drug: Ustekinumab; Drug: conventional treatment (glucocoticoid, immunosupressive drugs and/or mesalazine)

INTERVENTIONS:
Drug: Infliximab — A TNFα inhibitor in UC and CD treatment
  Other Names: IFX
Drug: Vedolizumab — An integrin receptor antagonist in UC and CD treatment
  Other Names: VDZ
  Groups: UC patients
Drug: Ustekinumab — An IL-12/IL-23 inhibitor in CD treatment
  Other Names: UST
  Groups: CD patients
Drug: conventional treatment (glucocoticoid, immunosupressive drugs and/or mesalazine) — Conventional treatment includes glucocoticoid, immunosupressive drugs and/or mesalazine. Immunosupressive drugs include azathioprine (AZA), methotrexate (MTX) and thalidomide (THA).
  Other Names: glucocoticoid, immunosupressive drugs, mesalazine (5-ASA)

SUMMARY:
Inflammatory bowel disease(IBD), including ulcerative colitis (UC) and Crohn's disease (CD), is characterized by chronic and recurrent nonspecific intestinal inflammation with high disability rate. During the past few decades, the prevalence of IBD is increasing, especially in developing countries, which brings great burden to patients themselves and medical insurance. Currently, biological medications such as TNFα inhibitors (infliximab, adalimumab, etc.), integrin receptor antagonist (vedolizumab) and interleukin 12/interleukin 23 inhibitor (ustekinumab) are commonly used in IBD treatment as well as traditional drugs such as glucocorticoid, immunosupressive agents and 5-Aminosalicylic Acid, and surgury. However, health-econimic analysis is lacking in Chinese IBD patients and more research is needed for making treatment choice.

Meanwhile, the etiology, disease progression and prognosis prediction has not totally been clarified. The efficacy prediction model of vedolizumab and infliximab has been analyzed, whose prediction markers include level of albumin, smoking, surgery history, fistula, etc. However, no model has included predictors concerning disease pathway or pharmacological pathway in patients accepting different therapy. So a model to predict IBD progression and prognosis concerning pharmacological pathway is going to be explored.

DETAILED DESCRIPTION:
The research is aimed at exploring the mode of IBD progression and predicting prognosis of different IBD patients so that treatment choice could be made to get better efficacy and decrease economic burden of patients and medical insurance. So blood and stool samples before and after treatment are collected to detect changes in gut microbiota and blood proteomics markers and explore the prediction model. Also, inflammatory bowel disease questionnaire (IBDQ) and EQ5D3L will be collected and cost-utility analysis will be conducted.

ELIGIBILITY:
Inclusion Criteria:

* be diagnosed CD or UC according to Chinese consensus on diagnosis and treatment in inflammatory bowel disease(2018, Beijing)
* willing to be followed up
* intend to be treated by biological agents (VDZ, IFX or UST) or conventional drugs (glucocoticoid±immunosupressive drugs±5-ASA)

Exclusion Criteria:

* with complex complications

Ages: 14 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This is a multicentered research and Chinese patients who meet the eligibility criteria will be enrolled. The medical centers are Peking Union Medical College Hospital, Beijing Chaoyang Hospital, Peking University Third Hospital, Beijing Shijingshan Hospital and the 7th Medical Center of PLA General Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-07-09 (Actual); Primary Completion 2023-09 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
endoscopic remission rate at week 12 | week 12 after treatment
  Endoscopic remission is defined as Mayo endoscopic subscore ≤1.

SECONDARY OUTCOMES:
clinical remission at week 0, 12 and 52 | week 0, week 12 and week 52 after treatment
  Clinical remission: defined as a Mayo score ≤2 and no individual subscore >1.

OTHER OUTCOMES:
side effect rate at week 0,12 and 52 | week 0, week 12 and week 52 after treatment
  side effect includes medication side effects, infection, reactivation of tuberculosis or hepatitis B, cancer, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Hong Yang, Doctor, Study Chair — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Torabi M, Bernstein CN, Yu BN, Wickramasinghe L, Blanchard JF, Singh H. Geographical Variation and Factors Associated With Inflammatory Bowel Disease in a Central Canadian Province. Inflamm Bowel Dis. 2020 Mar 4;26(4):581-590. doi: 10.1093/ibd/izz168. PMID 31504519
- [Background] Ng SC, Shi HY, Hamidi N, Underwood FE, Tang W, Benchimol EI, Panaccione R, Ghosh S, Wu JCY, Chan FKL, Sung JJY, Kaplan GG. Worldwide incidence and prevalence of inflammatory bowel disease in the 21st century: a systematic review of population-based studies. Lancet. 2017 Dec 23;390(10114):2769-2778. doi: 10.1016/S0140-6736(17)32448-0. Epub 2017 Oct 16. PMID 29050646
- [Background] Ouyang Q, Xue LY. Inflammatory bowel disease in the 21(st) century in China: turning challenges into opportunities. J Dig Dis. 2012 Apr;13(4):195-9. doi: 10.1111/j.1751-2980.2012.00579.x. PMID 22435503
- [Background] Ng SC, Kaplan GG, Tang W, Banerjee R, Adigopula B, Underwood FE, Tanyingoh D, Wei SC, Lin WC, Lin HH, Li J, Bell S, Niewiadomski O, Kamm MA, Zeng Z, Chen M, Hu P, Ong D, Ooi CJ, Ling KL, Miao Y, Miao J, Janaka de Silva H, Niriella M, Aniwan S, Limsrivilai J, Pisespongsa P, Wu K, Yang H, Ng KK, Yu HH, Wang Y, Ouyang Q, Abdullah M, Simadibrata M, Gunawan J, Hilmi I, Lee Goh K, Cao Q, Sheng H, Ong-Go A, Chong VH, Ching JYL, Wu JCY, Chan FKL, Sung JJY. Population Density and Risk of Inflammatory Bowel Disease: A Prospective Population-Based Study in 13 Countries or Regions in Asia-Pacific. Am J Gastroenterol. 2019 Jan;114(1):107-115. doi: 10.1038/s41395-018-0233-2. PMID 30177785
- [Background] Solberg IC, Lygren I, Jahnsen J, Aadland E, Hoie O, Cvancarova M, Bernklev T, Henriksen M, Sauar J, Vatn MH, Moum B; IBSEN Study Group. Clinical course during the first 10 years of ulcerative colitis: results from a population-based inception cohort (IBSEN Study). Scand J Gastroenterol. 2009;44(4):431-40. doi: 10.1080/00365520802600961. PMID 19101844
- [Background] Lv H, Jin M, Zhang H, Chen X, Wu M, Guo M, Zhou R, Wang Z, Yang H, Qian J. Increasing newly diagnosed inflammatory bowel disease and improving prognosis in China: a 30-year retrospective study from a single centre. BMC Gastroenterol. 2020 Nov 12;20(1):377. doi: 10.1186/s12876-020-01527-1. PMID 33183228
- [Background] Pillai N, Dusheiko M, Burnand B, Pittet V. A systematic review of cost-effectiveness studies comparing conventional, biological and surgical interventions for inflammatory bowel disease. PLoS One. 2017 Oct 3;12(10):e0185500. doi: 10.1371/journal.pone.0185500. eCollection 2017. PMID 28973005
- [Background] Jean L, Audrey M, Beauchemin C, Consortium OBOTI. Economic Evaluations of Treatments for Inflammatory Bowel Diseases: A Literature Review. Can J Gastroenterol Hepatol. 2018 Jun 13;2018:7439730. doi: 10.1155/2018/7439730. eCollection 2018. PMID 30009158